CLINICAL TRIAL: NCT00416325
Title: Phase I Multiple Dose Pharmacokinetic Study of Lycopene Delivered in a Well-Defined Food-Based Lycopene Delivery System (Tomato Paste-Oil Mixture) in Patients at Increased Risk for Developing Prostate Cancer
Brief Title: Lycopene in Preventing Prostate Cancer in Patients Who Are at High Risk of Developing Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: UIC-2000-0931; CDR0000467322 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

INTERVENTIONS:
Dietary Supplement: lycopene
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs or substances to keep cancer from forming, growing, or coming back. The use of lycopene, a substance found in tomatoes, may keep prostate cancer from forming in patients at high risk of developing prostate cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of lycopene in preventing prostate cancer in patients who are at high risk of developing prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the toxicity and safety of lycopene administered as a food-based delivery system as a chemoprevention agent in patients who are at a high risk of developing prostate cancer.
* Define the pharmacokinetics and tissue distribution in patients receiving this regimen.
* Characterize surrogate endpoint biomarkers (SEBs) in the peripheral blood, buccal mucosa, and the prostate itself, which will provide evidence of biological activity relevant to a chemoprevention effect.

  * Characterize the oxidative stress state of the individual by studies of DNA oxidation in the prostate and buccal mucosa, as well as DNA oxidation and lipid peroxidation within the peripheral blood.
  * Define the effects of lycopene through a food delivery system on prostate histology (prostatic intraepithelial neoplasia), markers of cellular proliferation [PCNA], and apoptosis in the prostate.
  * Evaluate the effects of lycopene on the serum levels of total prostate-specific antigen (PSA), free PSA, and PSA density.
* Provide the basic knowledge in reference to toxicity, pharmacokinetics, and SEBs needed to proceed to a large phase II or III lycopene study in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral lycopene in tomato paste and olive oil, once, twice, or three times daily for 3 months.

Cohorts of 6 patients receive escalating doses of lycopene until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients undergo buccal scrapings and blood collection periodically during study for pharmacokinetics and biomarker studies.

After completion of study treatment, patients are followed for 1 month.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Elevated prostate-specific antigen (PSA), meeting 1 of the following criteria:

  * PSA > 4.0 ng/mL for patients at any age
  * PSA > 2.0 ng/mL for patients 35 to 49 years of age
  * PSA rise (velocity) of > 0.75 ng/mL over the past year
* Has undergone a prostate biopsy* (following findings of elevated PSA) within the past 180 days that failed to reveal prostate cancer

  * Prostate intraepithelial neoplasia allowed NOTE: *At least 4 core biopsies are considered acceptable

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* WBC ≥ 3,000/mm^3
* Hemoglobin ≥ 11.0 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 125,000/mm^3
* No history of gastrointestinal malabsorption or other condition affecting drug absorption
* No history of food allergy to tomato-based products
* No history of any chronic medical condition that, in the judgment of the investigator, may pose threat or additional risk to the patient (including a current history of alcohol or drug abuse)
* No active history of cancer or other illnesses that, in the opinion of the investigator, could represent a threat to patient's life, including congestive heart failure or uncontrolled hypertension

PRIOR CONCURRENT THERAPY:

* No participation in any other experimental trial within the past 4 weeks
* No concurrent chronic use of nonsteroidal anti-inflammatory drugs
* No concurrent participation in another experimental trial
* No concurrent supplements (except multivitamins), including herbal and soy products

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Toxicity as measured by NCI CTC v2.0
Feasibility of daily consumption of prescribed volumes of the formulation
Serum lycopene levels, including other carotenoids and lipid soluble vitamins, at 1 and 3 months
Pharmacokinetics at 1 and 3 months
Tissue distribution of lycopene (oral mucosa and prostate tissue)
Modulation of surrogate endpoint biomarkers which include oxidative stress in blood, oral mucosa, and prostate tissue
Modulation of serum prostate-specific antigen
Cellular proliferation as measured by proliferating cell nuclear antigen (PCNA)
Apoptosis as measured by Terminal deoxynucleotidyl Transferase Biotin-dUTP Nick End Labeling in prostate tissue
Serum levels of insulin-like growth factor (IGF-1) and the modulation of prostate histology (prostatic intraepithelial neoplasia [PIN], when and if present)

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Rodvold, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Derived] Gann PH, Deaton RJ, Rueter EE, van Breemen RB, Nonn L, Macias V, Han M, Ananthanarayanan V. A Phase II Randomized Trial of Lycopene-Rich Tomato Extract Among Men with High-Grade Prostatic Intraepithelial Neoplasia. Nutr Cancer. 2015;67(7):1104-12. doi: 10.1080/01635581.2015.1075560. PMID 26422197